CLINICAL TRIAL: NCT03143725
Title: Open-label Study to Compare the Bioavailability of an Oral Wet Granulation Tablet of GLPG1972 Relative to an Oral Solution and to an Oral Direct Compression Tablet After Single-dose Intake in Healthy Subjects, and to Evaluate the Effect of Food on the Bioavailability of an Oral Wet Granulation Tablet.
Brief Title: Study to Compare Bioavailability of GLPG1972 Given as 2 Different Tablet Formulations Versus an Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1972-CL-105
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): GLPG1972 oral solution after overnight fast
  Interventions: Drug: GLPG1972
- Treatment B (Experimental): GLPG1972 oral DC tablet after breakfast
  Interventions: Drug: GLPG1972
- Treatment C (Experimental): GLPG1972 oral WG tablet after overnight fast
  Interventions: Drug: GLPG1972
- Treatment D (Experimental): GLPG1972 oral WG tablet after breakfast
  Interventions: Drug: GLPG1972

INTERVENTIONS:
Drug: GLPG1972 — Oral administration of GLPG1972 in four different treatment conditions (Treatments A throug D)

SUMMARY:
This study is a Phase I, randomized, open-label, cross-over study with 4 single-dose treatments of GLPG1972 to compare the bioavailability of the oral wet granulation (WG) tablet relative to an oral solution and to the oral direct compression (DC) tablet after single dose intake in healthy male subjects and to evaluate the effect of food on the bioavailability of the WG oral tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 and 50 years of age, inclusive,
2. A body mass index (BMI) between 18-30 kg/m², inclusive, weight of at least 50 kg.
3. Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and laboratory findings.
4. Discontinuation of all medications except occasional paracetamol at least 2 weeks or 5 half-lives prior to the first study drug administration.
5. Non-smokers and not using any nicotine-containing products.
6. Negative urine drug screen and alcohol breath test.
7. Current sexually active male agrees to use adequate contraception
8. Willing to consume a non-vegetarian high-fat and high-calorie breakfast
9. Able and willing to sign the ICF

Exclusion Criteria:

1. Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug
2. Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or any history of hepatitis from any cause with the exception of hepatitis A.
3. History of or a current immunosuppressive condition
4. Symptoms of clinically significant illness in the 3 months before the initial study drug administration.
5. History of malignancy within the past 5 years
6. Clinically relevant abnormalities detected on ECG regarding either rhythm or conduction (e.g. QTcF >450 msec, or a known long QT syndrome).
7. Presence of abnormal liver function
8. Renal function with an estimated creatinine clearance <80 ml/min based on the Cockcroft-Gault formula.
9. Presence of any condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
10. Clinically relevant abnormalities detected on "vital signs"
11. Dietary requirements precluding participation.
12. Significant blood loss including blood donation or had a transfusion of any blood product within 12 weeks
13. Hemoglobin level <7.5 mmol/L (12 g/dL).
14. Active drug or alcohol abuse within 2 years prior to the initial study drug administration.
15. Current (2 weeks before screening) and planned uninterrupted consumption of large quantities (> 6 cups) of coffee
16. Administration of an injectable drug within 30 days prior to the initial study drug administration.
17. Concurrent participation, or participation in a drug/device study within 8 weeks or 5 half-lives of the drug or within 6 months for biologicals
18. Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the maximum observed plasma concentration of GLPG1972 after single oral doses | on day 1 pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 and 48 hours post doses
  Determine bioavailability of GLPG1972 by assessing PK parameters
Assessment of plasma concentration of GLPG1972 24hrs post-dose after single oral doses | At 24 hours post dose
  Determine bioavailability of GLPG1972 by assessing PK parameters
Assessment of time to achieve the maximal plasma concentration of GLPG1972 after single oral doses | on day 1 pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 and 48 hours post doses
  Determine bioavailability of GLPG1972 by assessing PK parameters
Assessment of the last quantifiable plasma concentration of GLPG1972 after single oral doses | on day 1 pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 and 48 hours post doses
  Determine bioavailability of GLPG1972 by assessing PK parameters

SECONDARY OUTCOMES:
the number of subjects with adverse events | at screening, pre-dose at date 1 and post-dose at 24 and 48 hours
  To assess safety and tolerability of GLPG1972 given orally
the number of subjects with abnormal vital signs | at screening, pre-dose at date 1 and post-dose at 24 and 48 hours
  To assess safety and tolerability of GLPG1972 given orally
the number of subjects with abnormal ECG | at screening, pre-dose at date 1 and post-dose at 24 and 48 hours
  To assess safety and tolerability of GLPG1972 given orally
the number of subjects with abnormal laboratory assessments | at screening, pre-dose at date 1 and post-dose at 24 and 48 hours
  To assess safety and tolerability of GLPG1972 given orally

CONTACTS AND LOCATIONS:
Overall Officials: Ann Fieuw, MD MSc, Study Director — Galapagos NV
Locations (1):
- SGS Belgium Life Sciences, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided